CLINICAL TRIAL: NCT07369297
Title: EVALUATION OF ELECTRICAL AND THERMAL PULP SENSORY THRESHOLDS AND MASSETER INHIBITORY REFLEX RESPONSES IN PATIENTS WITH DIABETIC POLYNEUROPATHY
Brief Title: PULP SENSIBILITY AND MASSETER INHIBITORY REFLEX IN DIABETIC POLYNEUROPATHY
Status: Not yet recruiting | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: E.224974
Record Dates: First submitted 2026-01-07; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Polyneuropathy; Healthy Individuals (Controls)
Keywords: Diabetic Polyneuropathy; Electrical Pulp Test; Cold Test; Masseter Inhibitory Reflex
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Mild Diabetic Polyneuropathy: The severity of diabetic polyneuropathy will be determined based on nerve conduction studies performed by the Department of Neurology. Participants will be classified into mild or severe diabetic polyneuropathy groups according to standardized nerve conduction parameters, including sensory and motor nerve conduction velocities, amplitudes, and latencies. These classifications will be made by an experienced neurologist, and group allocation will be based on objective electrophysiological findings rather than subjective symptoms.
  Interventions will be performed in the following order: thermal (cold test), electric pulp test, and masseter inhibitory reflex recording.
- Severe Diabetic Polyneuropathy: The severity of diabetic polyneuropathy will be determined based on nerve conduction studies performed by the Department of Neurology. Participants will be classified into mild or severe diabetic polyneuropathy groups according to standardized nerve conduction parameters, including sensory and motor nerve conduction velocities, amplitudes, and latencies. These classifications will be made by an experienced neurologist, and group allocation will be based on objective electrophysiological findings rather than subjective symptoms. Interventions will be performed in the following order: thermal (cold test), electric pulp test, and masseter inhibitory reflex recording.
- Healthy Controls Group: The healthy control group will consist of individuals with no history of diabetes mellitus, peripheral neuropathy, or any other systemic or neurological disease. Control participants will have no history of chemotherapy, chronic pain disorders, or conditions known to affect peripheral nerve function. Individuals using medications that may influence sensory perception or nerve conduction within the last 24 hours will be excluded.
  Healthy controls will undergo the same standardized examination protocol as the diabetic polyneuropathy groups, including thermal (cold) testing, electric pulp testing, and masseter inhibitory reflex (MIR) recording, performed in the same fixed order. The same tooth selection criteria will be applied, and all procedures will be conducted under identical conditions to allow reliable comparison between groups.

SUMMARY:
Accurate evaluation of dental pulp health is essential to avoid unnecessary endodontic treatments. In routine dental practice, pulp sensibility is commonly assessed using electric pulp testing and thermal (cold) testing. However, these tests depend on patient perception and may be influenced by various factors such as systemic diseases, nerve damage, anxiety, trauma, or medication use.

Diabetic polyneuropathy is a common complication of diabetes mellitus and may alter peripheral nerve function, potentially affecting dental pulp sensibility test responses. This clinical study aims to evaluate how the severity of diabetic polyneuropathy influences dental pulp sensibility responses and masseter inhibitory reflex (MIR) parameters. The MIR is an objective neurophysiological reflex that allows quantitative assessment of trigeminal nerve function.

In this study, individuals with mild diabetic polyneuropathy, severe diabetic polyneuropathy, and healthy controls will be evaluated. All participants will undergo electric pulp testing, cold testing, and MIR measurements using standardized protocols.

The primary hypothesis of this study is that increasing severity of diabetic polyneuropathy leads to reduced dental pulp sensibility responses and altered MIR parameters compared to healthy individuals. It is further hypothesized that conventional pulp sensibility tests may produce false-negative results in patients with advanced neuropathy.

The findings of this study are expected to contribute to more accurate endodontic diagnosis and improved understanding of orofacial neurophysiological changes in diabetic patients.

DETAILED DESCRIPTION:
Accurate assessment of dental pulp health is fundamental for correct endodontic diagnosis and for preventing unnecessary or inappropriate treatment decisions. In routine dental practice, pulp sensibility is commonly evaluated using electric pulp testing (EPT) and thermal (cold) testing. These methods primarily assess neural response rather than true pulp vitality and rely on patient perception, which makes them inherently subjective.

Several factors may influence pulp sensibility test outcomes, including systemic diseases affecting peripheral nerves, such as diabetic polyneuropathy, as well as trauma, anxiety levels, medication use, and metabolic disease duration. Diabetic polyneuropathy is a frequent complication of diabetes mellitus and is characterized by progressive sensory nerve dysfunction. This condition may alter trigeminal nerve conduction and pain perception, potentially leading to altered or reduced responses in conventional pulp sensibility tests and increasing the risk of false-negative results.

The masseter inhibitory reflex (MIR) is a well-established neurophysiological reflex mediated by trigeminal afferent and efferent pathways and can be objectively recorded using electromyography. Unlike conventional pulp tests, MIR provides quantitative and objective information about orofacial sensory and motor nerve function. However, the relationship between diabetic polyneuropathy severity, dental pulp sensibility responses, and MIR parameters has not been sufficiently investigated.

The aim of this clinical study is to evaluate the effect of diabetic polyneuropathy severity on dental pulp sensibility responses and masseter inhibitory reflex parameters. Individuals diagnosed with diabetic polyneuropathy who presented to the Department of Neurology at Bezmialem Vakıf University will be included and categorized into mild and severe neuropathy groups based on neurological evaluation. A healthy control group without systemic or neurological disease will also be included for comparison.

A total of 108 participants aged between 25 and 65 years will be enrolled. Demographic and clinical data including age, sex, duration of diabetes, presence of comorbid systemic diseases other than diabetes, and medication use within the last 24 hours will be recorded for all participants.

Dental pulp sensibility tests will be performed on the maxillary central incisor. The selected tooth must be free of caries or present only with small, non-extensive restorations, must not have undergone root canal treatment, and must show no clinical or radiographic signs of periapical pathology or periodontal disease. Teeth with extensive caries, restorations, periodontal pathology, or previous endodontic treatment will be excluded.

Thermal sensibility will be assessed using a cold test, and both the time to initial sensation and the duration of sensation decay will be recorded.

Electric pulp testing will be performed using a standardized protocol, and the response threshold will be recorded as a numerical value on a scale ranging from 0 to 64. All pulp sensibility tests will be conducted under standardized conditions, and patient responses will be documented.

Masseter inhibitory reflex recordings will be obtained using electromyography. Electrical stimulation will be applied to the maxillary central incisor using a sterile needle electrode. Surface electrodes will be placed according to standardized neurophysiological protocols to record MIR responses. Participants may experience brief and mild transient sensations during stimulation. All procedures will be explained in detail prior to testing, and participants will be informed that they may request termination of the procedure at any time. If a participant expresses discomfort or wishes to stop, all procedures will be immediately discontinued.

The primary hypothesis of this study is that increasing severity of diabetic polyneuropathy is associated with decreased dental pulp sensibility responses and altered MIR parameters compared to healthy controls. It is further hypothesized that conventional pulp sensibility tests may yield false-negative responses in individuals with advanced neuropathy, whereas MIR measurements will provide objective evidence of altered orofacial nerve function.

Statistical analysis will be performed using appropriate statistical software. Descriptive statistics will be calculated for all variables. Normality of data distribution will be assessed using the Shapiro-Wilk test. Group comparisons will be conducted using one-way analysis of variance (ANOVA) or Kruskal-Wallis test, depending on data distribution. Post hoc analyses will be performed where appropriate. Associations between neuropathy severity, pulp sensibility parameters, and MIR measurements will be evaluated using correlation and regression analyses. A p-value of <0.05 will be considered statistically significant.

The results of this clinical study are expected to improve understanding of the impact of diabetic polyneuropathy on dental pulp sensibility testing and to support the use of neurophysiological assessment methods as complementary tools in endodontic diagnosis. By identifying limitations of conventional pulp tests in diabetic patients, this study aims to contribute to more accurate diagnostic decision-making and improved patient care.

ELIGIBILITY:
Inclusion Criteria:

Ability to understand the study procedures and provide written informed consent.

For diabetic polyneuropathy groups:

* Diagnosis of diabetic polyneuropathy confirmed by a neurologist
* Neuropathy severity (mild or severe) determined by nerve conduction studies

For healthy control group:

* No history of diabetes mellitus
* No history of peripheral neuropathy or neurological disease

Presence of at least one maxillary central incisor suitable for testing, defined as:

* No previous root canal treatment
* No extensive caries
* No clinical or radiographic signs of periapical pathology
* No periodontal disease affecting the selected tooth

Exclusion Criteria:

* History of chemotherapy, head and neck radiotherapy, or systemic conditions known to affect peripheral nerve function (other than diabetic polyneuropathy in the patient groups)
* Presence of acute or chronic orofacial pain disorders
* Use of medications within the last 24 hours that may affect sensory perception or nerve conduction (e.g., analgesics, sedatives, neuroactive drugs)
* History of trauma to the maxillary central incisor or surrounding tissues
* Extensive restorations, fractures, caries, or periodontal pathology involving the selected tooth
* Pregnancy or breastfeeding
* Inability to tolerate study procedures or refusal to continue participation at any point

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be selected from adult patients attending the Departments of Neurology and Endodontics at Bezmialem Vakif University. The study population will include individuals diagnosed with type 2 diabetes mellitus with mild and severe diabetic neuropathy who have been evaluated in the Neurology Department, as well as systemically healthy control subjects. Participants will be recruited from patients referred from the Neurology Department and from individuals presenting for routine dental examination at the university dental clinic.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Electrical Pulp Testing Threshold | The total duration of the EPT procedure is expected to be approximately 2-3 minutes per participant, including tooth isolation, probe placement, gradual increase of electrical stimulus intensity, and recording of the response threshold.
  Electric pulp sensibility will be evaluated using a standardized electric pulp test (EPT) performed on the maxillary central incisor. The tooth will be isolated and dried, and a conductive medium will be applied to ensure proper electrical contact. The EPT probe will be placed on the mid-facial surface of the tooth, and electrical stimulus intensity will be gradually increased according to the manufacturer's instructions. Participants will be instructed to indicate the first sensation perceived during stimulation. The stimulus will be stopped immediately upon participant response. The response threshold will be recorded as a numerical value on a standardized scale ranging from 0 to 64. The test will be repeated after a short recovery period if necessary to confirm reproducibility.

SECONDARY OUTCOMES:
Time to First Sensation During Thermal (cold) Pulp Sensibility Test | The thermal (cold) pulp sensibility test will require approximately 2-3 minutes, including tooth isolation, application of the cold stimulus, and recording of response times.
  Thermal (cold) pulp sensibility will be assessed using a standardized cold test performed on the maxillary central incisor. The tooth will be isolated and dried, and a cold stimulus will be applied to the mid-facial surface using a cotton pellet sprayed with refrigerant (e.g., 1,1,1,2-tetrafluoroethane). The stimulus will be maintained until the participant reports the first sensation. The test will be repeated after an appropriate recovery period to avoid sensitization. The time to first sensation will be recorded in seconds (s).
Time to Disappearance of Sensation After Thermal (cold) Stimulus Removal | The thermal (cold) pulp sensibility test will require approximately 2-3 minutes, including tooth isolation, application of the cold stimulus, and recording of response times.
  Using the same standardized cold test protocol, thermal (cold) pulp sensibility will be assessed on the maxillary central incisor. The tooth will be isolated and dried, and a cold stimulus will be applied to the mid-facial surface using a cotton pellet sprayed with refrigerant (e.g., 1,1,1,2-tetrafluoroethane). After the stimulus is removed, the time from removal of the cold stimulus to complete disappearance of the sensation will be recorded in seconds (s) to assess pulp sensibility recovery characteristics.
Masseter Inhibitory Reflex Latency | The total duration of MIR recording, including electrode placement, calibration, and electromyographic data acquisition, is expected to be approximately 10-15 minutes per participant.
  The masseter inhibitory reflex (MIR) will be recorded using electromyography to objectively assess trigeminal nerve function. Participants will be seated in a comfortable position, and electromyographic electrodes will be placed according to standardized neurophysiological protocols. Electrical stimulation will be delivered to the maxillary central incisor using a sterile needle electrode.
  The stimulation intensity will be set at 120% of the individual electric pulp test (EPT) sensory threshold. During stimulation, electromyographic activity of the masseter muscle will be recorded, and the latency of the silent periods (SP1 and SP2) will be measured in milliseconds (ms).
Masseter Inhibitory Reflex Silent Period Duration | The total duration of MIR recording, including electrode placement, calibration, and electromyographic data acquisition, is expected to be approximately 10-15 minutes per participant.
  Using a standardized electromyographic recording protocol, the masseter inhibitory reflex will be recorded to assess trigeminal nerve function. Participants will be seated in a comfortable position, and surface electromyographic electrodes will be placed over the masseter muscle according to established neurophysiological guidelines. Electrical stimulation will be delivered to the maxillary central incisor using a sterile needle electrode.
  The stimulation intensity will be set at 120% of the individual electric pulp test (EPT) sensory threshold. Following stimulation, the duration of the silent periods (SP1 and SP2) will be measured in milliseconds (ms) to assess inhibitory trigeminal reflex function.

DOCUMENTS (1):
  • Informed Consent Form (2025-12-31): https://cdn.clinicaltrials.gov/large-docs/97/NCT07369297/ICF_000.pdf